CLINICAL TRIAL: NCT04405141
Title: The Relationship Between Vitamin D Level and Lower Urinary Tract Symptoms in Women
Brief Title: Uroflowmetry Results and Vitamin D Levels
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sibel Ocak Serin, Principal investigator, Umraniye Education and Research Hospital
Other Study IDs: UmraniyeERH
Record Dates: First submitted 2020-05-09; First posted 2020-05-28 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Lower Urinary Tract Symptoms; Vitamin D Deficiency; Calcium Deficiency
Keywords: Lower Urinary Tract Symptoms; Vitamin D Deficiency; Calcium Deficiency
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to evaluate the relationship between LUTS and vitamin D with uroflowmetry parameters in female patients. They found no relation between vitamin D levels and LUTS in respect to uroflowmetry. However, in low vitamin D patients, Ca is related with urologic problems. The investigators believe that there is a need for studies emphasizing serum Ca levels in addition to vitamin D levels in patients with LUTS.

DETAILED DESCRIPTION:
This retrospective cohort study included 186 female patients who admitted to LUTS. Demographic characteristics, medical history, calcium (Ca) and vitamin D including laboratory studies and uroflowmetry results as maximum urine flow rate (Qmax), average urine flow rate (Qav), and voided volume (V) were recorded. Patients were divided into two groups according to age (18-50 and ≥51) and vitamin D levels (<20 and ≥20).

Laboratory parameters, uroflowmetry results, were compared between groups.

The study was approved by the local ethics committee (approval#22/06/2018-09.29-54132726-000-14136). The study was conducted in accordance to the Helsinki Declaration and Good Clinical Practices Guidelines.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of low urinary tract symptom

Exclusion Criteria:

Urinary tract infection, Diabetes mellitus, Neurological disorder, Pregnancy Stone disease Other urinary system disorders.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Because females are more related to low urinary tract symptoms.
Study Population: Female patients with low urinary tract symptoms.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Uroflowmetry Results | 12 months
  There was no significant relationship between age, creatinine, Qmax, Qav, V and vitamin D level (P>0.05).

SECONDARY OUTCOMES:
Vitamin D Levels | 12 months
  The mean D vitamin level was 21.19ng/ml. D vitamin was <20 ng/ml in %55.9 patients. There was no difference in the levels according to the age of all patients.